CLINICAL TRIAL: NCT07229183
Title: Midwifery Students' Family Planning Counseling and Material Development Skills and the Effectiveness of Standardized Patient Simulation and Peer Simulation
Brief Title: Family Planning Counseling and Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Döndü BATKIN ERTÜRK, Assistant professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TOKAT05
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Educational Problems
Keywords: midwifery student; family planning; peer simulation; standardized patient simulation; education material

STUDY DESIGN:
Intervention Model Description: Participants were divided into three groups: standardized patient simulation, peer simulation, and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standardized Patient Group (Experimental): Trained with SP in simulation sessions
  Interventions: Behavioral: Standardized patient simulation practice
- Peer Simulation Group (Experimental): Trained with a peer in simulation sessions
  Interventions: Behavioral: Peer Simulation practice
- Control Group (No Intervention): No intervention was made

INTERVENTIONS:
Behavioral: Standardized patient simulation practice — Creating family planning scenarios Preparing educational materials Identifying and training standardized patients on the scenarios Providing family planning counseling with standardized patients in simulation sessions accompanied by educational materials
  Arms: Standardized Patient Group
Behavioral: Peer Simulation practice — Creating family planning scenarios Preparing educational materials Identifying and training peers on the scenarios Providing family planning counseling in simulation sessions with peers using educational materials
  Arms: Peer Simulation Group

SUMMARY:
The purpose of this experimental study is to investigate the effects of standardized patient simulation and peer simulation on midwifery students' family planning counseling and material development skills.

The main questions it aims to answer are:

Do standardized patient simulation and peer simulation training affect midwifery students' family planning counseling skills?

Do standardized patient simulation and peer simulation training affect midwifery students' material development skills?

The researchers will compare simulation groups with a control group to determine whether simulation training improves midwifery students' family planning counseling and material development skills.

Participants:

For the peer simulation, three volunteer second-year midwifery students will portray a peer in the client role.

Three volunteer undergraduate/master's students with prior theater training will portray a standardized patient in the client role.

The control group, without receiving simulation training, will prepare educational material on general family planning counseling after the simulation sessions and present this material to their peers in a classroom setting as a counseling practice.

Simulation groups will complete the State/Trait Anxiety Inventory before simulation and family planning counseling, and the control group will complete the State/Trait Anxiety Inventory before family planning counseling.

DETAILED DESCRIPTION:
The goal of family planning services is to improve pregnancy planning and spacing and to prevent unintended pregnancies. They enable individuals to achieve desired birth spacing and family size and contribute to improved health outcomes for children, women, and families. According to the World Health Organization (2014) and the United Nations (2014), all couples and individuals have the right to freely and responsibly decide on the number, spacing, and timing of their children and to have the information and tools necessary to do so. Family planning provides multifaceted benefits for women and their families.

It is unique among health interventions in terms of its breadth of health, development, and economic benefits, including reducing maternal and child mortality, empowering women and girls, and increasing environmental sustainability. Midwives play a crucial role in improving maternal and infant health and providing family planning and reproductive health services.

Family planning relies, in part, on the communication skills and attitudes of healthcare providers involved in counseling. A study demonstrated that a client-centered approach to family planning counseling, which fosters shared decision-making, builds trust, and explores client preferences, increases satisfaction and retention. Another study suggests that midwifery students need more practical training in contraception and sexual health.

The use of printed educational materials is recommended to supplement and reinforce health information commonly delivered orally, thereby increasing the effectiveness of health education. According to Bernier, written educational materials offer a number of advantages, including message consistency, reusability, portability, distribution flexibility, information retention, and cost-effectiveness of production and updating. Healthcare professionals should provide written health education materials designed according to best-practice principles in written health education material design and focused on the healthy/ill individual. Health education materials are only effective if they are read, understood, and remembered by healthy/ill individuals.

By writing their own educational materials, health educators can adapt content to the policies, procedures, and equipment of their respective institutions, create answers to frequently asked questions by healthy and sick individuals, emphasize points deemed particularly important by healthcare professionals, and reinforce specific verbal instructions that clarify difficult concepts and address specific healthy and sick needs.

In this context, enhancing midwifery students' material development skills is crucial.

Standardized patients are individuals who have received special training to accurately convey a patient's story so accurately that even experienced healthcare professionals cannot distinguish them from real patients. By embodying all the physical and psychological characteristics of real patients, they provide students with a holistic understanding of patient care. These individuals are frequently used in health sciences education to promote the development of communication skills and other core competencies.

They can consistently represent a wide variety of scenarios. Issues such as high cost, standardized patient training, and other limitations limit the use of standardized patients in health education. A potential alternative to standardized patients is to have students role-play the patient. Peer simulation is an advanced form of role-playing in which students are trained to role-play clinical scenarios for their peers. While there are studies examining the impact of simulation on improving family planning counseling, no studies have been found comparing the effectiveness of standardized patient simulation with peer simulation.

In addition, this study focuses on the ability to prepare educational materials on the subject as well as family planning counseling.

ELIGIBILITY:
Inclusion Criteria:

* Students taking the course for the first time
* Students who agree to participate in the research
* Students who continue the theoretical part of the course

Exclusion Criteria:

- Students who did not attend simulation sessions

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
State/Trait Anxiety Inventory | Pre-simulation (Baseline) and Pre-family planning counseling
  1. Not at all,
  2. A little,
  3. A lot, and 4) Completely
General Counseling Evaluation Form in Family Planning | Throughout family planning counseling-10 minutes
  "1 = needs improvement" (steps are implemented incorrectly or skipped),
  "2 = adequate" (steps are implemented correctly and in the correct order, but progress from step to step is not smooth),
  "3 = mastered" (steps are implemented correctly and in the correct order, and progress is smooth from step to step)
Patient Education Material Evaluation Tool | Pre-family planning counseling- 5 minutes
  Disagree = 0 points Agree = 1 point No Rating

CONTACTS AND LOCATIONS:
Overall Officials: Döndü BATKIN ERTÜRK, Assist.Prof., Principal Investigator — Tokat Gaziosmanpaşa University
Locations (1):
- Tokat Gaziosmanpaşa Üniversitesi, Tokat Province, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma KA, Zangmo R, Kumari A, Roy KK, Bharti J. Family planning and abortion services in COVID 19 pandemic. Taiwan J Obstet Gynecol. 2020 Nov;59(6):808-811. doi: 10.1016/j.tjog.2020.09.005. Epub 2020 Sep 10. PMID 33218393
- [Background] Ensuring Human Rights in the Provision of Contraceptive Information and Services: Guidance and Recommendations. Geneva: World Health Organization; 2014. Available from http://www.ncbi.nlm.nih.gov/books/NBK195054/ PMID 24696891
- [Background] United Nations Population Fund (2023) Human Rights-Based Approach To Family Planning, UNFPA Support Tool. Available at: https://www.unfpa.org/sites/default/files/pub-pdf/UNFPA-HRBAtoFP-SupportTool-v231207.pdf Accessed:18 March 2025
- [Background] Şimşek Çetinkaya, Ş., Gümüş Çalış, G., Kıbrıs, Ş., & Topal, M. (2024). Effectiveness of virtual patient simulation versus peer simulation in family planning training in midwifery students: a comparative educational intervention. Interactive Learning Environments, 32(3), 942-951.
- [Background] Li Q, Rimon JG, Ahmed S. Capitalising on shared goals for family planning: a concordance assessment of two global initiatives using longitudinal statistical models. BMJ Open. 2019 Nov 12;9(11):e031425. doi: 10.1136/bmjopen-2019-031425. PMID 31722946
- [Background] Inurreta-Díaz, M., Morales-Gual, Y. M., Aguilar-Vargas, E., Álvarez-Baeza, A., Magriñá-Lizama, J. S., Cetina-Sauri, G., & Méndez-Domínguez, N. (2021). Family-Planning counselling simulation for medical students: An exploratory educational intervention. Educación médica, 22, 271-276.
- [Background] Schivone GB, Glish LL. Contraceptive counseling for continuation and satisfaction. Curr Opin Obstet Gynecol. 2017 Dec;29(6):443-448. doi: 10.1097/GCO.0000000000000408. PMID 28938374
- [Background] Walker SH, Davis G. Knowledge and reported confidence of final year midwifery students regarding giving advice on contraception and sexual health. Midwifery. 2014 May;30(5):e169-76. doi: 10.1016/j.midw.2014.02.002. Epub 2014 Feb 25. PMID 24661469
- [Background] Sim, K. H. (2011). Tips for creating effective health education materials. The Journal of Korean Diabetes, 12(2), 99-103.
- [Background] Hoffmann T, Worrall L. Designing effective written health education materials: considerations for health professionals. Disabil Rehabil. 2004 Oct 7;26(19):1166-73. doi: 10.1080/09638280410001724816. PMID 15371031
- [Background] Hainsworth D. & Keyes K. Chapter 12: Instructional materials. In: Bastable SB. (ed.) Nurse as educator: Principles of teaching and learning for nursing practice, Fifth Edition Jones & Bartlett Learning; 2019. p 505-48.
- [Background] Ghorbani B, Jackson AC, Dehghan-Nayeri N, Bahramnezhad F. Standardized patients' experience of participating in medical students' education: a qualitative content analysis. BMC Med Educ. 2024 May 28;24(1):586. doi: 10.1186/s12909-024-05531-x. PMID 38807118